CLINICAL TRIAL: NCT03068767
Title: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Brief Title: The Relationship Between Vitamin D and Hepatitis B Virus Replication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, Chia-Chi Wang, Department of Gastroenterology, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TZ-105
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Results first posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Vitamin D and Hepatitis B Virus
Keywords: HBV DNA, qHBsAg
MeSH Terms: conditions — Hepatitis B | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: Group 1: vitamin D supplement Group 2: controls

ARMS (2):
- Vitamin D group (Experimental): Patients receiving vitamin D supplement (2000 IU/day) for 2 months
  Interventions: Dietary Supplement: Vitamin D
- Control group (No Intervention): Patients without receiving vitamin D supplement

INTERVENTIONS:
Dietary Supplement: Vitamin D
  Arms: Vitamin D group

SUMMARY:
149 HBV carriers with inadequate serum vitamin D levels were randomized to two groups: one is supplied with vitamin D and another without as controls. The markers of HBV replication were compared before and after treatment.

DETAILED DESCRIPTION:
This is a randomized case-control trial. A total of 149 HBV carriers with inadequate vitamin D (< 30 ng/mL) level were enrolled. They were randomly divided to two groups: one group receiving vitamin D supplement (1600 IU/day) for 2 months and another group as controls. The serum vitamin D, HBV DNA and qHBsAg levels were measured at baseline and after vitamin D supplement. Whether HBV DNA and qHBsAg have significant change after vitamin D supplement can be determined.

ELIGIBILITY:
Inclusion Criteria:

* >20 y/o, HBV carrier
* serum vitamin D < 30ng/ml

Exclusion Criteria:

* Other known causes of hepatitis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2016-09; Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Chi CC Wang, Master, Principal Investigator — Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Locations (1):
- Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Chronic HBV patients receiving regular 6-month surveillance in the outpatient clinic of Taipei Tzu Chi Hospital were invited to join the study from August 2017 to September 2018.
Pre-assignment Details: All had positive hepatitis B surface antigen (HBsAg) for more than 6 months. Those with positive anti-hepatitis C virus (HCV) antibody, other known causes of chronic hepatitis or receiving antiviral treatment currently were excluded. Those who had HBsAg loss, undetectable HBV DNA and adequate vitamin D level (≥30 ng/mL) were excluded.
Groups:
- Vitamin D Group: Patients receiving vitamin D supplement (2000 IU/day) for 2 months
  Vitamin D
Period: Overall Study
Arm/Group | Vitamin D Group | Control Group
Started | 75 (from August 2017 to September 2018) | 74 (from August 2017 to September 2018)
Completed | 65 (December 2018) | 71 (December 2018)
Not Completed | 10 | 3
Not completed — Lost to Follow-up | 7 | 3
Not completed — Protocol Violation | 3 | 0

BASELINE CHARACTERISTICS:
Population: Those who had HBsAg loss, undetectable HBV DNA and adequate vitamin D level (≥30 ng/mL) were excluded. The eligible subjects were randomized into two groups by using the computer random distribution.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D Group | Control Group | Total
Number analyzed (Participants) | 75 | 74 | 149
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 65 | 68 | 133
  >=65 years | 10 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Those who had HBsAg loss, undetectable HBV DNA and adequate vitamin D level (≥30 ng/mL) were excluded. The eligible subjects were randomized into two groups by using the computer random distribution.
  years | 51.85 (10.88) | 51.28 (8.86) | 51.61 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Those who had HBsAg loss, undetectable HBV DNA and adequate vitamin D level (≥30 ng/mL) were excluded. The eligible subjects were randomized into two groups by using the computer random distribution.
  Participants
    Female | 43 | 40 | 83
    Male | 32 | 34 | 66
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Dynamic Change of HBV DNA
Description: the serum HBV DNA levels were measured in CH-B patients before and after 2-month vitamin D supplement
Time Frame: baseline, after 2-month vitamin D supplement
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Vitamin D Group | Control Group
Number analyzed (Participants) | 75 | 74
IU/mL | 3.15 (1.14) | 3.14 (1.36)

2. Primary Outcome: The Change of Serum qHBsAg (IU/mL)
Description: The serum qHBsAg levels were measured before and after 2-month vitamin D supplement
Time Frame: baseline, after 2-month vitamin D supplement
Population: Levels of qHBsAg before and after 2 months of vitamin D treatment or follow-up were compared between these two groups.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Vitamin D Group | Control Group
Number analyzed (Participants) | 75 | 74
IU/mL | 2.19 (1.03) | 2.4 (1.11)

ADVERSE EVENTS:
Time Frame: 2 months
Description: Death: 0% Serious adverse event: 0% adverse event: 6%
Groups:
- Vitamin D Group: Patients receiving vitamin D supplement (2000 IU/day) for 2 months
  Vitamin D
  No serious adverse events noted.
- Control Group: Patients without receiving vitamin D supplement
  No serious adverse events noted.
Arm/Group | Vitamin D Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/74
Other Adverse Events (participants affected / at risk) | 3/75 | 6/74
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D Group (N=75) | Control Group (N=74)
tearing (Eye disorders) | 0 (0) | 1 (1) — increased tear
urine occult blood positive (Renal and urinary disorders) | 1 (1) | 0 (0) — Positive urine occult blood in urinalysis
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — feel difficulty in breathing
skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — skin rash over legs
sneezing (Ear and labyrinth disorders) | 0 (0) | 2 (2) — sneezing
acid reflux (Gastrointestinal disorders) | 0 (0) | 1 (1) — sometimes acid reflux
leg soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — leg soreness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT03068767/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT03068767/SAP_001.pdf